CLINICAL TRIAL: NCT01145729
Title: Clinical Response to Biomarker Documentation of Child Secondhand Smoke Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institutes of Health (NIH) (NIH)
Responsible Party: Anne Joseph, University of Minnesota
Organization: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-03

CONDITIONS: Biomarker Feedback; Smoking Cessation; Secondhand Smoke Exposure; Provider Behavior
Keywords: Biomarker feedback; Smoking cessation; Childhood secondhand smoke exposure
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biomarker feedback (Active Comparator): Biomarkers of tobacco exposure (laboratory values) delivered to health care provider
  Interventions: Behavioral: Biomarker Feedback
- Usual care (general counseling) (Placebo Comparator): Brochure about pesticides, lead, SHS
  Interventions: Behavioral: Biomarker Feedback

INTERVENTIONS:
Behavioral: Biomarker Feedback — Providing providers biomarker feedback on childhood secondhand smoke exposure

SUMMARY:
1. To do formative work with healthcare providers, clinic staff and parents to develop a protocol for a clinic system to routinely collect blood from children at risk of SHS exposure conduct laboratory testing for tobacco toxicants, document exposure in the electronic medical record (EMR) and incorporate the biomarker feedback into a parental smoking treatment plan.
2. To pilot test effects of a clinic system to screen children at risk of SHS exposure with laboratory testing for tobacco toxicants on provider delivery of tobacco treatment services (primary outcome).
3. To pilot test effects of a clinic system to screen children at risk of SHS exposure with laboratory testing for tobacco toxicants on parent smoking behavior (participation in smoking cessation treatment, smoking cessation and implementation of smoking restrictions).

DETAILED DESCRIPTION:
ABSTRACT Smoking and secondhand smoke (SHS) are responsible for nearly a half-million preventable deaths in the United States every year. Parent(s) who stop smoking incur health benefits, model non-smoking (and quitting) to children and stop exposure to SHS in the home, car and other locations. National initiatives from the American Academy of Pediatrics and the American Academy of Family Physicians urge healthcare providers to screen children for a history of SHS exposure and to recommend that parents stop smoking and restrict smoking at home, but compliance with these guidelines is poor and more than 25% of children in the U.S. continue to be involuntarily exposed to SHS in the home. Effective systems are needed to increase parental smoking cessation and implement home smoking restrictions. We propose preliminary studies to evaluate a novel intervention to accomplish these objectives. We hypothesize that a clinic system that routinely measures and reports levels of tobacco toxicants (tobacco-specific carcinogens, nicotine and cotinine) found in the urine of children exposed to SHS will 1) increase provider delivery of tobacco treatment, 2) increase parental participation in tobacco treatment, 3) increase parental smoking cessation and 4) reduce childhood exposure to secondhand smoke. We propose formative work among healthcare providers and parents to develop the intervention and to pilot test the effects of the intervention on providers and parents. We will conduct focus groups among staff to identify training needs, develop methods to integrate the intervention with office practice and assess barriers to implementation. We will also conduct focus groups among parents to assess willingness to provide urine specimens, optimal feedback format and reactions to biomarker data. Results from focus groups will be used to develop the experimental treatment protocol. We will test the intervention in a two-group randomized pilot study in the University of Minnesota Primary Care Clinic. We will recruit 80 children age 0-12 with a parent who smokes. We will provide brief behavioral counseling in healthy lifestyle options to all parents. One provider team will implement the experimental intervention in 40 parent-child pairs and the other team will serve as the control. Children who see providers in the experimental group will provide a urine sample to test for nitrosamines (a tobacco-specific carcinogen), nicotine and cotinine. We will communicate laboratory results to providers using the electronic medical record and incorporate these results in parental tobacco counseling designed to promote smoking cessation and home smoking restrictions. The primary outcome will be provider delivery of smoking cessation treatment. We will also measure effects on parental engagement in treatment, smoking cessation and institution of home smoking restrictions in both the experimental and control groups. The research team brings extensive experience with novel tobacco interventions, health services research and biomarker assessment to the project. Routine documentation of tobacco toxicants in children's urine has potential to dramatically alter clinical care for families at risk from smoking.

ELIGIBILITY:
Inclusion Criteria:

* 12M or 24M well-visit
* Scheduled to a lead test
* Current smoker

Exclusion Criteria:

* Cannot speak English
* No phone

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Provider Delivery of Tobacco Treatment Services | 12 weeks
  Whether or not biomarker feedback testing of secondhand smoke will prompt providers to deliver tobacco treatment services

SECONDARY OUTCOMES:
Parent Smoking Behavior | 12 weeks
  Whether giving parents biomarker feedback on childhood exposure to secondhand smoke will lead to participation in smoking cessation treatment, smoking cessation and implementation of smoking restrictions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Department of Medicine, Minneapolis, Minnesota, United States